CLINICAL TRIAL: NCT05961280
Title: Upstaging and Lymph Node Metastasis Rate in Patients With Ductal Carcinoma in Situ Who Received Mastectomy Regarding the Necessary of Sentinel Lymph Node Biopsy
Brief Title: Selective Omission of Sentinel Lymph Node Biopsy in Mastectomy for Ductal Carcinoma in Situ: Identifying Eligible Candidates
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Joon Jeong, Professor, Gangnam Severance Hospital
Other Study IDs: 3-2023-0026
Record Dates: First submitted 2023-07-06; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Ductal Carcinoma in Situ
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Mastectomy; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DCIS Mastectomy: Patients who undergo mastectomy with sentinel lymph node biopsy for DCIS at biopsy
  Interventions: Procedure: Mastectomy with sentinel lymph node biopsy

INTERVENTIONS:
Procedure: Mastectomy with sentinel lymph node biopsy

SUMMARY:
This study aimed to assess the prevalence of upgrade to invasive breast cancer and axillary lymph node metastasis in patients who were diagnosed with DCIS on biopsy and subsequently underwent mastectomy with axillary surgery to establish the need for SLNB. Furthermore, we explored the clinicopathologic features related to the upgrade to invasive breast cancer and axillary lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Women diagnosed with DCIS in preoperative biopsy samples obtained by core needle biopsy, vacuum-assisted breast biopsy, or excisional biopsy
2. Women underwent curative surgery for DCIS

Exclusion Criteria:

1. Patients who received breast-conserving surgery
2. Patients who had concurrent contralateral invasive breast cancer
3. Patients who were in case of ipsilateral breast tumor recurrence
4. Patients whose invasiveness was uncertain in the biopsy samples

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent mastectomy with sentinel lymphnode biopsy for DCIS.
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Axillary lymph node metastasis rate | up to 2 weeks after surgery
  Our primary objective was to identify the axillary lymph node metastasis rate in patients with DCIS at diagnosis who underwent mastectomy with axillary surgery.